CLINICAL TRIAL: NCT04394247
Title: Patient Characteristics, Treatment Patterns, and Clinical Outcomes in Patients Diagnosed With HR+/HER2- Advanced/Metastatic Breast Cancer Receiving Palbociclib + Aromatase Inhibitor (AI) Combination Therapy as First-Line Treatment
Brief Title: Patient Characteristics, Treatment Patterns, and Clinical Outcomes in Patients Diagnosed With HR+/HER2 Advanced/Metastatic Breast Cancer on Palbociclib + Aromatase Inhibitor (AI) Combination Therapy
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A5481155
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer Patients: HR + /HER2- Advanced/Metastatic Breast Cancer patients in U.S.A

SUMMARY:
The study is designed to describe patient characteristics, treatment patterns, and clinical effectiveness outcomes in patients diagnosed with HR+/HER2- A/MBC who received palbociclib combination therapy with AI as first-line treatment in the US community oncology setting.

ELIGIBILITY:
Inclusion Criteria:

* Female or male sex.
* Diagnosis (confirmed by clinical review) of A/MBC, defined as breast cancer at stage IIIB, stage IIIC, stage IV or identified as having distant metastasis.
* Age ≥18 years at A/MBC diagnosis.
* Initiated palbociclib in combination with an AI as first-line therapy after A/MBC diagnosis on or after 03 February 2015 through 31 July 2019. Note that the date of the start of the inclusion period reflects the month of palbociclib US FDA approval.
* Evidence of ER or PR positive disease, or absence of any indication of ER and PR negative disease closest to A/MBC diagnosis (ie, patients are eligible without affirmative indication of ER/PR+ status as long as ER/PR- indication is not present).
* Evidence of HER2 negative disease, or absence of any indication of HER2 positive disease closest to A/MBC diagnosis (ie, patients are eligible without affirmative indication of HER2- status as long as HER2+ indication is not present).

Exclusion Criteria:

* Enrollment in an interventional clinical trial for A/MBC during the study observation period.
* Evidence of prior treatment with any CDK4/6 inhibitor in the adjuvant setting.
* Evidence of another primary cancer within 3 years prior to the initial line containing palbociclib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients 18 years or older, diagnosed with HR+/HER2- A/MBC who initiated palbociclib combination therapy with AI as the first-line therapy on or after 03 February 2015 up to and including 31 July 2019.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Syapse, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Law JW, Mitra D, Kaplan HG, Alfred T, Brufsky AM, Emir B, McCracken H, Liu X, Broome RG, Zhang C, DiCristo C, Chen C. Real-World Treatment Patterns and Clinical Effectiveness of Palbociclib Plus an Aromatase Inhibitor as First-Line Therapy in Advanced/Metastatic Breast Cancer: Analysis from the US Syapse Learning Health Network. Curr Oncol. 2022 Feb 12;29(2):1047-1061. doi: 10.3390/curroncol29020089. PMID 35200588
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A5481155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who received palbociclib with aromatase inhibitor(AI) as first-line therapy on or after 03 February 2015 through 31 July 2019 were observed retrospectively; data cutoff was 01 February 2020, resulting in a minimum potential 6-month follow-up period. The data was abstracted from charts during a 6 month period of time from 30 June 2020 to 31 December 2020.
Groups:
- Palbociclib With Aromatase Inhibitor: Participants with advanced/metastatic breast cancer (A/MBC), hormone receptor (HR) positive and human epidermal growth factor receptor 2 (HER2) negative disease, received palbociclib capsule orally once daily with AI as first-line therapy were observed retrospectively during the study. The data of these participants were studied in this observational study.
Period: Overall Study
Arm/Group | Palbociclib With Aromatase Inhibitor
Started | 242
Completed | 242
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all participants who met following criteria: 1) Diagnosis of A/MBC; 2) Aged >=18 years at A/MBC diagnosis; 3) Initiated palbociclib in combination with AI as first-line therapy after A/MBC diagnosis on or after 03 February 2015 through 31 July 2019; 4) Evidence of estrogen receptor(ER) or progesterone receptor(PR) positive disease and HER2 negative disease or absence of any indication of ER and PR negative disease and HER2 positive disease closest to A/MBC diagnosis.
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Age, Continuous [Mean (Standard Deviation); unit: Years] — Age at initial diagnosis
  Years | 60.39 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 238
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15
  Not Hispanic or Latino | 225
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 10
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 29
  White | 196
  More than one race | 0
  Unknown or Not Reported | 6
Year of Initial Diagnoses [Median (Full Range); unit: Years] | 2016 [1987 to 2019]
Year of A/MBC Diagnoses [Median (Full Range); unit: Year] | 2017 [2011 to 2019]
Age at A/MBC Diagnosis [Mean (Standard Deviation); unit: Years] | 64.68 (12.22)
Age at Death [Number; unit: Percentage of participants]
  Less than (<) 50 years | 1.7
  Between 50-64 years | 9.9
  Between 65-74 years | 5.4
  Greater than or equal to (>=) 75 years | 8.7
  Missing | 74.0
Insurance Carrier at A/MBC Diagnosis [Number; unit: Percentage of Participants] — Here, percentage of participants with their insurance status at A/MBC diagnosis as medicare/medicaid, commercial, not stated in participant record and none categories were reported.
  Percentage of Participants
    Medicare/Medicaid | 61.6
    Commercial | 28.5
    Not Stated in Participant Record | 8.7
    None | 1.2
Menopausal Status at A/MBC Diagnosis [Number; unit: Percentage of participants] — Menopausal status at time of A/MBC diagnosis that included pre-menopausal, post-menopausal, peri-menopausal, not stated in participant record and not applicable were reported.
  Percentage of participants
    Post-menopausal | 85.5
    Pre-menopausal | 9.9
    Peri-menopausal | 0.8
    Not Stated in Participant Record | 2.1
    Not Applicable | 1.7
Region of Residence at A/MBC Diagnosis [Number; unit: Percentage of participants] — Here, percentage of participants with region of residence at A/MBC diagnosis as northeast, south, north central and west were reported.
  Percentage of participants
    Northeast | 0.4
    South | 4.1
    North Central | 95.0
    West | 0.4
Stage at Initial Breast Cancer Diagnosis [Number; unit: Percentage of participants] — Percentage of participants stages 0, I, IA, II, IIA, IIB, III, IIIA, IIIB, IIIC, IV, not stated in participant record were reported. American Joint Committee on Cancer staging, 0=noninvasive ductal carcinoma in situ; I=tumor <=2centimeters(cm), no lymph node; IA= <2cm,no spread; II= 2-5cm, spread to lymph nodes; IIA= 1-3 lymph nodes with or without <2cm/2-5cm,no lymph node; IIB=2-5cm, nearby lymph nodes/>5cm, no lymph node; III=spread to lymph nodes; IIIA=any size, 4-9 lymph nodes; IIIB=spread to chest wall; IIIC=any size,10 or more lymph nodes; IV(metastatic)=any size, spread to other organs.
  Percentage of participants
    0 | 0.8
    I | 2.9
    IA | 1.2
    II | 6.6
    IIA | 8.3
    IIB | 9.5
    III | 2.5
    IIIA | 5.0
    IIIB | 0.4
    IIIC | 0.8
    IV | 55.4
    Not Stated in Participant Record | 7
Percentage of Participants With Histology Type [Number; unit: Percentage of participants] — Here, percentage of participants were reported according to type of histology as invasive ductal carcinoma, invasive lobular carcinoma, invasive mixed (ductal and lobular), ductal carcinoma in situ (DCIS) and other.
  Percentage of participants
    Invasive Ductal Carcinoma | 56.6
    Invasive Lobular Carcinoma | 22.3
    Invasive Mixed (ductal and lobular) | 4.5
    DCIS | 0.8
    Other | 15.7
Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: Percentage of participants] — Percentage of participants with their ECOG performance status at baseline were recorded and reported. ECOG performance status measurement at baseline included scores from 0 to 3 where, 0= fully active, no performance restrictions; 1= strenuous physical activity restricted, fully ambulatory and able to carry out light work; 2= capable of all self-care but unable to carry out any work activities, up and about greater than (>) 50 percent (%) of waking hours; 3= capable of only limited self-care; confined to bed or chair >50% of waking hours.
  Percentage of participants
    ECOG- 0 | 23.6
    ECOG- 1 | 24.0
    ECOG- 1-2 | 0.4
    ECOG- 2 | 8.3
    ECOG- 3 | 3.3
    ECOG- Not Stated in Participant Record | 40
Percentage of Participants With Any Prior Surgery [Number; unit: Percentage of participants] — Here, percentage of participants were classified according to any prior surgery as Yes or No.
  Percentage of participants
    Yes | 52.5
    No | 47.5
Percentage of Participants With Types of Surgery [Number; unit: Percentage of participants] — Here, percentage of participants were classified according to types of surgery as breast conserving surgery and mastectomy.
  Percentage of participants
    Breast Conserving Surgery | 20.2
    Mastectomy | 32.2
Percentage of Participants With Radiation Therapy [Number; unit: Percentage of participants] — Here, percentage of participants were classified according to radiation therapy as Yes or No.
  Percentage of participants
    Yes | 32.6
    No | 67.4
Percentage of Participants With Radiation Therapy Sites [Number; unit: Percentage of participants] — Here, percentage of participants with radiation therapy sites as chest wall, regional lymph nodes; partial breast; whole breast; whole breast, regional lymph nodes; chest wall and unknown were reported.
  Percentage of participants
    Chest Wall, Regional Lymph Nodes | 7.4
    Partial Breast | 0.8
    Whole Breast | 7.4
    Whole Breast, Regional Lymph Nodes | 5.0
    Chest Wall | 5.0
    Unknown (site not known) | 7.4
Percentage of Participants With Comorbid Disease Burden [Number; unit: Percentage of participants] — Comorbidities at baseline included hypertension, diabetes, renal disease, chronic pulmonary disease, anemia, congestive heart failure, cardiac arrhythmia, peripheral vascular disease, rheumatic disease, cerebrovascular disease, dementia, myocardial infarction, liver disease, not stated in participant record and none of the above categories.
  Percentage of participants
    Hypertension | 48.8
    Diabetes | 21.9
    Renal Disease | 9.1
    Chronic Pulmonary Disease | 5.8
    Anemia | 4.5
    Congestive Heart Failure | 4.1
    Cardiac Arrhythmias | 2.9
    Peripheral Vascular Disease | 1.2
    Rheumatic Disease | 1.2
    Cerebrovascular Disease | 0.8
    Dementia | 0.8
    Myocardial Infarction | 0.8
    Liver Disease | 0.4
    Not Stated in Participant Record | 1.2
    None of the Above | 36.8
Percentage of Participants With Charlson Comorbidity Index Score [Number; unit: Percentage of participants] — Charlson comorbidity index (CCI) scored the cumulative severity of a participant's comorbidities. Total score ranged from 0 to 9. A score of zero indicated that no comorbidities were found. The higher the score, the more likely the cumulative severity of a participant's comorbidities. CCI was calculated based on the presence of 17 charlson comorbidities at A/MBC.
  Percentage of participants
    0 | 65.3
    1 | 19.4
    2 | 9.1
    3 | 3.7
    4+ | 2.5
Percentage of Participants With Sites of Distant Metastasis [Number; unit: Percentage of participants] — Here, percentage of participants with sites of distant metastasis as bone (bone only or in addition to other sites), bone only, chest wall, central nervous system (CNS), contralateral breast, distant lymph node(s), visceral sites, liver, lung, peritoneum, pleural nodules, malignant pleural effusion, skin, ovary, adrenal, bone marrow, colon, omentum, soft tissue, stomach, other specify were reported.
  Percentage of participants
    Bone (Bone only or in addition to other sites) | 83.1
    Bone Only | 50.8
    Chest Wall | 0.0
    CNS | 2.5
    Contralateral Breast | 0.8
    Distant Lymph Node (s) | 18.6
    Visceral Sites | 32.2
    Liver | 9.9
    Lung | 21.5
    Peritoneum | 2.1
    Pleural Nodules | 5
    Malignant Pleural Effusion | 10.3
    Skin | 3.7
    Ovary | 0.4
    Adrenal | 1.7
    Bone Marrow | 1.7
    Colon | 0.8
    Omentum | 0.4
    Soft Tissue | 2.5
    Stomach | 1.2
    Other: Specify | 7.4
Percentage of Participants With Number of Metastatic Sites [Number; unit: Percentage of participants] — Here, percentage of participants were reported according to number of metastatic sites.
  Percentage of participants
    1 | 60.7
    2 | 18.6
    >=3 | 20.2
    Participant is Not Metastatic | 0.4
Percentage of Participants With Disease Burden at Metastatic Sites in Liver [Number; unit: Percentage of participants] — Here, percentage of participants with disease burden at metastatic sites in liver were reported as single lesion, multiple lesions, unknown number of lesions and no metastases at site.
  Percentage of participants
    Single Lesion | 3.3
    Multiple Lesions | 5.8
    Unknown Number of Lesions | 0.8
    No Metastases at Site | 90.1
Percentage of Participants With Disease Burden at Metastatic Sites in Lung [Number; unit: Percentage of participants] — Here, percentage of participants with disease burden at metastatic sites in lung were reported as single lung, bilateral lungs, unknown single vs bilateral status and no metastases at site.
  Percentage of participants
    Single Lung | 5.4
    Bilateral Lungs | 13.2
    Unknown Single vs Bilateral Status | 2.9
    No Metastases at Site | 78.5
Percentage of Participants With Disease Burden at Metastatic Sites in Bone [Number; unit: Percentage of participants] — Here, percentage of participants with disease burden at metastatic sites in bone were reported as single site, multiple sites, unknown number of sites and no metastases at site.
  Percentage of participants
    Single Site | 16.9
    Multiple Sites | 64.5
    Unknown Number of Sites | 1.7
    No Metastases at Site | 16.9
Percentage of Participants With Time to Metastasis [Number; unit: Percentage of participants] — Time to metastasis was defined as months between initial and metastasis diagnoses. It was categorized into less than or equal to (<=)12 months, 13-24 months, 25-36 months and greater than (>)36 months. Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Percentage of participants
    <= 12 Months: number analyzed (Participants) | 105
    <= 12 Months | 5.7
    13-24 Months: number analyzed (Participants) | 105
    13-24 Months | 3.8
    25-36 Months: number analyzed (Participants) | 105
    25-36 Months | 8.6
    > 36 Months: number analyzed (Participants) | 105
    > 36 Months | 81.9
Percentage of Participants With HER2 and Estrogen Receptor (ER) or Progesterone Receptor (PR) Status [Number; unit: Percentage of participants] — Here, percentage of participants with HER2 and ER or PR status as positive (+), negative (-) and equivocal were reported.
  Percentage of participants
    HER2 Status: HER2 negative | 97.9
    HER2 Status: equivocal | 2.1
    Hormone Receptor Status: ER+ / PR+ | 79.8
    Hormone Receptor Status: ER+ / PR- | 18.6
    Hormone Receptor Status: ER+ / Not Applicable (NA) | 0.8
    Hormone Receptor Status: ER- / PR+ | 0.4
    Hormone Receptor Status: ER- / PR- | 0.4
Percentage of Participants With Breast Cancer Susceptibility Gene (BRCA) 1 or 2 Testing Status [Number; unit: Percentage of participants] — Here, percentage of participants were classified according to BRCA 1 or 2 testing status as Yes or No.
  Percentage of participants
    Yes | 19.0
    No | 81.0
Percentage of Participants With Modalities of Treatment Received Prior to A/MBC [Number; unit: Percentage of participants] — Neoadjuvant participants those who received modalities of treatment prior to A/MBC. It included chemotherapy, endocrine therapy, and targeted therapy for neoadjuvant participants. Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Percentage of participants
    Chemotherapy: number analyzed (Participants) | 99
    Chemotherapy | 12.1
    Endocrine Therapy: number analyzed (Participants) | 99
    Endocrine Therapy | 7.1
    Targeted Therapy: number analyzed (Participants) | 99
    Targeted Therapy | 1.0
Percentage of Participants With Endocrine Sensitivity and Endocrine Resistance [Number; unit: Percentage of participants] — Endocrine sensitivity: >=12 months without recurrence/progression after completion of endocrine therapy in the adjuvant setting. Primary endocrine resistance: relapse within 2 years of adjuvant endocrine therapy or progressive disease within 6 months of first-line endocrine therapy for metastatic breast cancer. Secondary endocrine resistance: relapse while on adjuvant endocrine therapy but after 2 years of treatment, relapse within 12 months of completing adjuvant endocrine therapy, or progressive disease >=6 months after starting endocrine therapy for metastatic breast cancer. Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Percentage of participants
    Endocrine Sensitivity: number analyzed (Participants) | 53
    Endocrine Sensitivity | 84.9
    Primary Endocrine Resistance | 28.5
    Secondary Endocrine Resistance | 45.5
Disease Free Interval [Median (Full Range); unit: Months] — Disease free interval was defined as months from the end of adjuvant therapy till the date of disease recurrence. Population: Here, number analyzed signifies participants evaluable for this baseline measure.
  Months
    number analyzed (Participants) | 105
    (all) | 64.00 [0 to 299.0]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Regimen Distribution
Description: Regimen medications were defined as systemic therapies included in line regimen based on synapse line of therapy algorithm. Treatment regimen distribution included: first-line regimen; palbociclib along with aromatase inhibitor and second-line regimen; CDK4/6 inhibitor plus endocrine and chemotherapy. Systemic anticancer treatment here refers to one or more sequential monotherapy or combination therapy regimens occurring within discrete lines of treatment, each ending with a disease progression.
Time Frame: From start of treatment to end of follow-up, up to a maximum of approximately 5 years
Population: Analysis population included all participants who met following criteria: 1) Diagnosis of A/MBC; 2) Aged >=18 years at A/MBC diagnosis; 3) Initiated palbociclib in combination with AI as first-line therapy after A/MBC diagnosis on or after 03 February 2015 through 31 July 2019; 4) Evidence of ER or PR positive disease and HER2 negative disease or absence of any indication of ER and PR negative disease and HER2 positive disease closest to A/MBC diagnosis.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Percentage of participants
  First-line regimen | 100
  Second-line regimen | 39.67

2. Primary Outcome: Percentage of Participants With Sequence of Treatment Lines
Description: Line of therapy was defined as line number (1; 2; 3; etc.) in the A/MBC setting assigned based on synapse line of therapy algorithm. Systemic anticancer treatment here refers to one or more sequential monotherapy or combination therapy regimens occurring within discrete lines of treatment, each ending with a disease progression.
Time Frame: From start of treatment to end of follow-up, up to a maximum of approximately 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Percentage of participants
  1 Line | 100
  2 Lines | 21.49
  3 Lines | 12.81
  4 Lines | 2.07
  5 Lines or more | 3.31

3. Primary Outcome: Percentage of Participants With Their Starting Dose and End Dose
Description: Percentage of participants with starting and end dose at 125 mg, 100 mg, 75 mg and unknown were reported.
Time Frame: From start of treatment to end of follow-up, up to a maximum of approximately 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Percentage of participants
  Starting Dose: 125 mg | 89.7
  Starting Dose: 100 mg | 7.4
  Starting Dose: 75 mg | 1.2
  Starting Dose: Unknown | 1.7
  End Dose: 125 mg | 60.7
  End Dose: 100 mg | 27.7
  End Dose: 75 mg | 9.9
  End Dose: Unknown | 1.7

4. Primary Outcome: Percentage of Participants With Type of Dose Adjustment
Description: In this outcome measure type of dose adjustments were recorded and reported. It included dose increase, decrease, no adjustment and unknown categories.
Time Frame: From start of treatment to end of follow-up, up to a maximum of approximately 5 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Percentage of participants
  Increase | 0.4
  Decrease | 31.0
  No adjustment | 66.9
  Unknown | 1.7

5. Primary Outcome: Percentage of Participants With Their Reason For Treatment Discontinuation
Description: Percentage of participants with discontinuation reason as progression, intolerance/toxicity, participant choice, treatment for other diseases, left health system, end of planned therapy, changes in insurance, death, hospice referral, physician choice, actionable mutation found, other/unknown were recorded and reported in this outcome measure.
Time Frame: From start of treatment to end of follow-up, up to a maximum of approximately 5 years
Population: Analysis population (AP) included all participants who met following criteria: 1) Diagnosis of A/MBC; 2) Aged >=18 years at A/MBC diagnosis; 3) Initiated palbociclib in combination with AI as first-line therapy after A/MBC diagnosis on or after 03 February 2015 through 31 July 2019; 4) Evidence of ER or PR positive disease and HER2 negative disease or absence of any indication of ER and PR negative disease and HER2 positive disease closest to A/MBC diagnosis.
Measure: Number; unit: Percentage of participants
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Percentage of participants
  Progression | 26.4
  Intolerance/toxicity | 14.9
  Participant Choice | 2.5
  Treatment for Other Diseases | 2.5
  Left Health System | 0
  End of Planned Therapy | 2.1
  Changes in Insurance | 1.2
  Death | 1.2
  Hospice Referral | 1.2
  Physician Choice | 0.8
  Actionable Mutation Found | 0.4
  Other/Unknown | 2.9

6. Primary Outcome: Time to Dose Adjustment
Description: Time to dose adjustment (TTDA) was defined as the time from the start of palbociclib and AI treatment until the date of treatment dose adjustment.
Time Frame: From start of treatment till treatment dose adjustment, up to a maximum of approximately 5 years
Population: AP: all participants who met following criteria: 1)Diagnosis of A/MBC;2)Aged >=18years at A/MBC diagnosis;3)Initiated palbociclib in combination with AI as first-line therapy after A/MBC diagnosis on/after 03 February 2015-31 July 2019;4)Evidence of ER/PR positive disease and HER2 negative disease/absence of any indication of ER and PR negative disease and HER2 positive disease closest to A/MBC diagnosis. Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Days
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 76
Days | 55.0 [1.000 to 1435]

7. Primary Outcome: Probability of Real-World Progression-Free Survival (rwPFS) at Month 3
Description: Probability of being event free (event defined as disease progression [PD] or death due to any cause) at 3 months. rwPFS was defined as the extent of time from the start of palbociclib and AI treatment until disease progression, date of death prior to initiation of the 2nd line treatment. Participants who were not indicated to be deceased at the time of analysis were censored for rwPFS analysis at the date of initiation of the 2nd line treatment, date of last contact or the end of study period whichever occurred first. Probability of participants with rwPFS at 3 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 3 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being event free | 0.95 [0.92 to 0.97]

8. Primary Outcome: Probability of Real-World Progression-Free Survival (rwPFS) at Month 6
Description: Probability of being event free (event defined as PD or death due to any cause) at 6 months. rwPFS was defined as the extent of time from the start of palbociclib and AI treatment until disease progression, date of death prior to initiation of the 2nd line treatment. Participants who were not indicated to be deceased at the time of analysis were censored for rwPFS analysis at the date of initiation of the 2nd line treatment, date of last contact or the end of study period whichever occurred first. Probability of participants with rwPFS at 6 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 6 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being event free | 0.84 [0.8 to 0.89]

9. Primary Outcome: Probability of Real-World Progression-Free Survival (rwPFS) at Month 12
Description: Probability of being event free (event defined as PD or death due to any cause) at 12 months. rwPFS was defined as the extent of time from the start of palbociclib and AI treatment until disease progression, date of death prior to initiation of the 2nd line treatment. Participants who were not indicated to be deceased at the time of analysis were censored for rwPFS analysis at the date of initiation of the 2nd line treatment, date of last contact or the end of study period whichever occurred first. Probability of participants with rwPFS at 12 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 12 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being event free | 0.75 [0.7 to 0.81]

10. Primary Outcome: Probability of Real-World Progression-Free Survival (rwPFS) at Month 18
Description: Probability of being event free (event defined as PD or death due to any cause) at 18 months. rwPFS was defined as the extent of time from the start of palbociclib and AI treatment until disease progression, date of death prior to initiation of the 2nd line treatment. Participants who were not indicated to be deceased at the time of analysis were censored for rwPFS analysis at the date of initiation of the 2nd line treatment, date of last contact or the end of study period whichever occurred first. Probability of participants with rwPFS at 18 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 18 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being event free | 0.66 [0.59 to 0.72]

11. Primary Outcome: Probability of Real-World Progression-Free Survival (rwPFS) at Month 24
Description: Probability of being event free (event defined as PD or death due to any cause) at 24 months. rwPFS was defined as the extent of time from the start of palbociclib and AI treatment until disease progression, date of death prior to initiation of the 2nd line treatment. Participants who were not indicated to be deceased at the time of analysis were censored for rwPFS analysis at the date of initiation of the 2nd line treatment, date of last contact or the end of study period whichever occurred first. Probability of participants with rwPFS at 24 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 24 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being event free | 0.59 [0.53 to 0.67]

12. Primary Outcome: Probability of Real-World Progression-Free Survival (rwPFS) at Month 30
Description: Probability of being event free (event defined as PD or death due to any cause) at 30 months. rwPFS was defined as the extent of time from the start of palbociclib and AI treatment until disease progression, date of death prior to initiation of the 2nd line treatment. Participants who were not indicated to be deceased at the time of analysis were censored for rwPFS analysis at the date of initiation of the 2nd line treatment, date of last contact or the end of study period whichever occurred first. Probability of participants with rwPFS at 30 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 30 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being event free | 0.53 [0.46 to 0.61]

13. Primary Outcome: Probability of Real-World Progression-Free Survival (rwPFS) at Month 36
Description: Probability of being event free (event defined as PD or death due to any cause) at 36 months. rwPFS was defined as the extent of time from the start of palbociclib and AI treatment until disease progression, date of death prior to initiation of the 2nd line treatment. Participants who were not indicated to be deceased at the time of analysis were censored for rwPFS analysis at the date of initiation of the 2nd line treatment, date of last contact or the end of study period whichever occurred first. Probability of participants with rwPFS at 36 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 36 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being event free
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being event free | 0.48 [0.4 to 0.57]

14. Primary Outcome: Probability of Real-World Overall Survival (rwOS) at Month 3
Description: rwOS was defined as the time from the start of palbociclib and AI treatment until the date of death, date of last contact or the end of study period. Participants who were not indicated to be deceased at the time of analysis were censored for rwOS analysis at the date of last contact or the end of study period whichever occurred first. Probability of participants with rwOS at 3 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 3 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being alive
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being alive | 0.99 [0.97 to 1]

15. Primary Outcome: Probability of Real-World Overall Survival (rwOS) at Month 6
Description: rwOS was defined as the time from the start of palbociclib and AI treatment until the date of death, date of last contact or the end of study period. Participants who were not indicated to be deceased at the time of analysis were censored for rwOS analysis at the date of last contact or the end of study period whichever occurred first. Probability of participants with rwOS at 6 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 6 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being alive
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being alive | 0.97 [0.94 to 0.99]

16. Primary Outcome: Probability of Real-World Overall Survival (rwOS) at Month 12
Description: rwOS was defined as the time from the start of palbociclib and AI treatment until the date of death, date of last contact or the end of study period. Participants who were not indicated to be deceased at the time of analysis were censored for rwOS analysis at the date of last contact or the end of study period whichever occurred first. Probability of participants with rwOS at 12 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 12 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being alive
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being alive | 0.9 [0.87 to 0.94]

17. Primary Outcome: Probability of Real-World Overall Survival (rwOS) at Month 18
Description: rwOS was defined as the time from the start of palbociclib and AI treatment until the date of death, date of last contact or the end of study period. Participants who were not indicated to be deceased at the time of analysis were censored for rwOS analysis at the date of last contact or the end of study period whichever occurred first. Probability of participants with rwOS at 18 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 18 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being alive
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being alive | 0.84 [0.79 to 0.89]

18. Primary Outcome: Probability of Real-World Overall Survival (rwOS) at Month 24
Description: rwOS was defined as the time from the start of palbociclib and AI treatment until the date of death, date of last contact or the end of study period. Participants who were not indicated to be deceased at the time of analysis were censored for rwOS analysis at the date of last contact or the end of study period whichever occurred first. Probability of participants with rwOS at 24 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 24 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being alive
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being alive | 0.78 [0.72 to 0.84]

19. Primary Outcome: Probability of Real-World Overall Survival (rwOS) at Month 30
Description: rwOS was defined as the time from the start of palbociclib and AI treatment until the date of death, date of last contact or the end of study period. Participants who were not indicated to be deceased at the time of analysis were censored for rwOS analysis at the date of last contact or the end of study period whichever occurred first. Probability of participants with rwOS at 30 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 30 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being alive
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being alive | 0.73 [0.67 to 0.8]

20. Primary Outcome: Probability of Real-World Overall Survival (rwOS) at Month 36
Description: rwOS was defined as the time from the start of palbociclib and AI treatment until the date of death, date of last contact or the end of study period. Participants who were not indicated to be deceased at the time of analysis were censored for rwOS analysis at the date of last contact or the end of study period whichever occurred first. Probability of participants with rwOS at 36 months were reported in this outcome measure. Analysis was performed using Kaplan-Meier method.
Time Frame: 36 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability of being alive
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability of being alive | 0.69 [0.62 to 0.77]

21. Primary Outcome: Probability of Participants Without First Line Treatment Discontinuation or Death at Month 3
Description: Probability of participants without first-line treatment discontinuation or death at month 3 were reported in this outcome measure. Real-world time to treatment discontinuation (rwTTD) was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date the participant discontinued first-line therapy or date of death. Participant alive and without first-line therapy discontinuation were censored at the earliest of last known use of first-line therapy or end of study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 3 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.93 [0.9 to 0.96]

22. Primary Outcome: Probability of Participants Without First Line Treatment Discontinuation or Death at Month 6
Description: Probability of participants without first-line treatment discontinuation or death at month 6 were reported in this outcome measure. rwTTD was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date the participant discontinued first-line therapy or date of death. Participant alive and without first-line therapy discontinuation were censored at the earliest of last known use of first-line therapy or end of study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 6 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.84 [0.8 to 0.89]

23. Primary Outcome: Probability of Participants Without First Line Treatment Discontinuation or Death at Month 12
Description: Probability of participants without first-line treatment discontinuation or death at month 12 were reported in this outcome measure. rwTTD was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date the participant discontinued first-line therapy or date of death. Participant alive and without first-line therapy discontinuation were censored at the earliest of last known use of first-line therapy or end of study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 12 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.67 [0.61 to 0.74]

24. Primary Outcome: Probability of Participants Without First Line Treatment Discontinuation or Death at Month 18
Description: Probability of participants without first-line treatment discontinuation or death at month 18 were reported in this outcome measure. rwTTD was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date the participant discontinued first-line therapy or date of death. Participant alive and without first-line therapy discontinuation were censored at the earliest of last known use of first-line therapy or end of study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 18 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.56 [0.5 to 0.63]

25. Primary Outcome: Probability of Participants Without First Line Treatment Discontinuation or Death at Month 24
Description: Probability of participants without first-line treatment discontinuation or death at month 24 were reported in this outcome measure. rwTTD was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date the participant discontinued first-line therapy or date of death. Participant alive and without first-line therapy discontinuation were censored at the earliest of last known use of first-line therapy or end of study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 24 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.49 [0.42 to 0.56]

26. Primary Outcome: Probability of Participants Without First Line Treatment Discontinuation or Death at Month 30
Description: Probability of participants without first-line treatment discontinuation or death at month 30 were reported in this outcome measure. rwTTD was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date the participant discontinued first-line therapy or date of death. Participant alive and without first-line therapy discontinuation were censored at the earliest of last known use of first-line therapy or end of study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 30 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.41 [0.34 to 0.48]

27. Primary Outcome: Probability of Participants Without First Line Treatment Discontinuation or Death at Month 36
Description: Probability of participants without first-line treatment discontinuation or death at month 36 were reported in this outcome measure. rwTTD was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date the participant discontinued first-line therapy or date of death. Participant alive and without first-line therapy discontinuation were censored at the earliest of last known use of first-line therapy or end of study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 36 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.36 [0.3 to 0.44]

28. Primary Outcome: Probability of Participants Without Subsequent Line of Therapy Initiation or Death at Month 3
Description: Probability of participants without subsequent line of therapy initiation or death at month 3 were reported in this outcome measure. Real-world time to next treatment (rwTTNT) was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent line of treatment, date of death, date of last contact or the end of study period. Participant alive and without subsequent line of therapy initiation were censored at the earliest of the following events: date of last contact or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 3 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.97 [0.96 to 0.99]

29. Primary Outcome: Probability of Participants Without Subsequent Line of Therapy Initiation or Death at Month 6
Description: Probability of participants without subsequent line of therapy initiation or death at month 6 were reported in this outcome measure. rwTTNT was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent line of treatment, date of death, date of last contact or the end of study period. Participant alive and without subsequent line of therapy initiation were censored at the earliest of the following events: date of last contact or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 6 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.89 [0.85 to 0.93]

30. Primary Outcome: Probability of Participants Without Subsequent Line of Therapy Initiation or Death at Month 12
Description: Probability of participants without subsequent line of therapy initiation or death at month 12 were reported in this outcome measure. rwTTNT was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent line of treatment, date of death, date of last contact or the end of study period. Participant alive and without subsequent line of therapy initiation were censored at the earliest of the following events: date of last contact or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 12 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.73 [0.68 to 0.79]

31. Primary Outcome: Probability of Participants Without Subsequent Line of Therapy Initiation or Death at Month 18
Description: Probability of participants without subsequent line of therapy initiation or death at month 18 were reported in this outcome measure. rwTTNT was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent line of treatment, date of death, date of last contact or the end of study period. Participant alive and without subsequent line of therapy initiation were censored at the earliest of the following events: date of last contact or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 18 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.62 [0.56 to 0.69]

32. Primary Outcome: Probability of Participants Without Subsequent Line of Therapy Initiation or Death at Month 24
Description: Probability of participants without subsequent line of therapy initiation or death at month 24 were reported in this outcome measure. rwTTNT was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent line of treatment, date of death, date of last contact or the end of study period. Participant alive and without subsequent line of therapy initiation were censored at the earliest of the following events: date of last contact or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 24 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.55 [0.49 to 0.63]

33. Primary Outcome: Probability of Participants Without Subsequent Line of Therapy Initiation or Death at Month 30
Description: Probability of participants without subsequent line of therapy initiation or death at month 30 were reported in this outcome measure. rwTTNT was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent line of treatment, date of death, date of last contact or the end of study period. Participant alive and without subsequent line of therapy initiation were censored at the earliest of the following events: date of last contact or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 30 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.47 [0.4 to 0.55]

34. Primary Outcome: Probability of Participants Without Subsequent Line of Therapy Initiation or Death at Month 36
Description: Probability of participants without subsequent line of therapy initiation or death at month 36 were reported in this outcome measure. rwTTNT was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent line of treatment, date of death, date of last contact or the end of study period. Participant alive and without subsequent line of therapy initiation were censored at the earliest of the following events: date of last contact or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 36 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.41 [0.34 to 0.5]

35. Primary Outcome: Probability of Participants Without Subsequent Chemotherapy or Death at Month 3
Description: Probability of participants without subsequent chemotherapy or death at month 3 were reported in this outcome measure. Real-world time to chemotherapy (rwTTC) was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent chemotherapy or date of death. Participant alive and without subsequent chemotherapy were censored at the earliest of the following events: date of last contact or end of the study period, whichever came later. Analysis was performed using Kaplan-Meier method.
Time Frame: 3 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.98 [0.97 to 1]

36. Primary Outcome: Probability of Participants Without Subsequent Chemotherapy or Death at Month 6
Description: Probability of participants without subsequent chemotherapy or death at month 6 were reported in this outcome measure. rwTTC was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent chemotherapy or date of death. Participant alive and without subsequent chemotherapy were censored at the earliest of the following events: date of last contact or end of the study period, whichever came later. Analysis was performed using Kaplan-Meier method.
Time Frame: 6 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.93 [0.9 to 0.97]

37. Primary Outcome: Probability of Participants Without Subsequent Chemotherapy or Death at Month 12
Description: Probability of participants without subsequent chemotherapy or death at month 12 were reported in this outcome measure. rwTTC was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent chemotherapy or date of death. Participant alive and without subsequent chemotherapy were censored at the earliest of the following events: date of last contact or end of the study period, whichever came later. Analysis was performed using Kaplan-Meier method.
Time Frame: 12 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.83 [0.78 to 0.88]

38. Primary Outcome: Probability of Participants Without Subsequent Chemotherapy or Death at Month 18
Description: Probability of participants without subsequent chemotherapy or death at month 18 were reported in this outcome measure. rwTTC was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent chemotherapy or date of death. Participant alive and without subsequent chemotherapy were censored at the earliest of the following events: date of last contact or end of the study period, whichever came later. Analysis was performed using Kaplan-Meier method.
Time Frame: 18 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.74 [0.68 to 0.8]

39. Primary Outcome: Probability of Participants Without Subsequent Chemotherapy or Death at Month 24
Description: Probability of participants without subsequent chemotherapy or death at month 24 were reported in this outcome measure. rwTTC was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent chemotherapy or date of death. Participant alive and without subsequent chemotherapy were censored at the earliest of the following events: date of last contact or end of the study period, whichever came later. Analysis was performed using Kaplan-Meier method.
Time Frame: 24 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.69 [0.63 to 0.76]

40. Primary Outcome: Probability of Participants Without Subsequent Chemotherapy or Death at Month 30
Description: Probability of participants without subsequent chemotherapy or death at month 30 were reported in this outcome measure. rwTTC was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent chemotherapy or date of death. Participant alive and without subsequent chemotherapy were censored at the earliest of the following events: date of last contact or end of the study period, whichever came later. Analysis was performed using Kaplan-Meier method.
Time Frame: 30 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.63 [0.56 to 0.71]

41. Primary Outcome: Probability of Participants Without Subsequent Chemotherapy or Death at Month 36
Description: Probability of participants without subsequent chemotherapy or death at month 36 were reported in this outcome measure. rwTTC was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: start of subsequent chemotherapy or date of death. Participant alive and without subsequent chemotherapy were censored at the earliest of the following events: date of last contact or end of the study period, whichever came later. Analysis was performed using Kaplan-Meier method.
Time Frame: 36 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.58 [0.5 to 0.66]

42. Primary Outcome: Probability of Participants Without a First Line Therapy Dose Adjustment at Month 3
Description: Probability of participants without a first-line therapy dose adjustment at month 3 were reported in this outcome measure. Real-world time to dose adjustment (rwTTDA) was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date of first-line treatment dose adjustment or discontinuation, date of death, date of last contact or the end of study period. Participant alive and without a first-line therapy dose adjustment were censored at the earliest of the following events: first-line discontinuation, death, date of last contact, or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 3 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.82 [0.77 to 0.87]

43. Primary Outcome: Probability of Participants Without a First Line Therapy Dose Adjustment at Month 6
Description: Probability of participants without a first-line therapy dose adjustment at month 6 were reported in this outcome measure. rwTTDA was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date of first-line treatment dose adjustment or discontinuation, date of death, date of last contact or the end of study period. Participant alive and without a first-line therapy dose adjustment were censored at the earliest of the following events: first-line discontinuation, death, date of last contact, or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 6 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.76 [0.71 to 0.82]

44. Primary Outcome: Probability of Participants Without a First Line Therapy Dose Adjustment at Month 12
Description: Probability of participants without a first-line therapy dose adjustment at month 12 were reported in this outcome measure. rwTTDA was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date of first-line treatment dose adjustment or discontinuation, date of death, date of last contact or the end of study period. Participant alive and without a first-line therapy dose adjustment were censored at the earliest of the following events: first-line discontinuation, death, date of last contact, or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 12 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.73 [0.67 to 0.79]

45. Primary Outcome: Probability of Participants Without a First Line Therapy Dose Adjustment at Month 18
Description: Probability of participants without a first-line therapy dose adjustment at month 18 were reported in this outcome measure. rwTTDA was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date of first-line treatment dose adjustment or discontinuation, date of death, date of last contact or the end of study period. Participant alive and without a first-line therapy dose adjustment were censored at the earliest of the following events: first-line discontinuation, death, date of last contact, or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 18 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.69 [0.63 to 0.76]

46. Primary Outcome: Probability of Participants Without a First Line Therapy Dose Adjustment at Month 24
Description: Probability of participants without a first-line therapy dose adjustment at month 24 were reported in this outcome measure. rwTTDA was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date of first-line treatment dose adjustment or discontinuation, date of death, date of last contact or the end of study period. Participant alive and without a first-line therapy dose adjustment were censored at the earliest of the following events: first-line discontinuation, death, date of last contact, or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 24 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.68 [0.62 to 0.74]

47. Primary Outcome: Probability of Participants Without a First Line Therapy Dose Adjustment at Month 30
Description: Probability of participants without a first-line therapy dose adjustment at month 30 were reported in this outcome measure. rwTTDA was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date of first-line treatment dose adjustment or discontinuation, date of death, date of last contact or the end of study period. Participant alive and without a first-line therapy dose adjustment were censored at the earliest of the following events: first-line discontinuation, death, date of last contact, or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 30 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.67 [0.6 to 0.74]

48. Primary Outcome: Probability of Participants Without a First Line Therapy Dose Adjustment at Month 36
Description: Probability of participants without a first-line therapy dose adjustment at month 36 were reported in this outcome measure. rwTTDA was defined as length of time from the start of first-line therapy with palbociclib plus an aromatase inhibitor to the earliest of one the following: date of first-line treatment dose adjustment or discontinuation, date of death, date of last contact or the end of study period. Participant alive and without a first-line therapy dose adjustment were censored at the earliest of the following events: first-line discontinuation, death, date of last contact, or end of the study period. Analysis was performed using Kaplan-Meier method.
Time Frame: 36 months after treatment initiation any time during 5 years of study period
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Palbociclib With Aromatase Inhibitor
Number analyzed (Participants) | 242
Probability | 0.65 [0.59 to 0.73]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: From start of treatment up to a maximum of approximately 5 years. Data for non-serious adverse events and serious adverse events (SAEs) were not collected and evaluated during the study; hence timeframe is not applicable for non-SAEs and SAEs
Description: Due to non-interventional nature of the study, data for non-SAEs and SAEs were not collected.
Arm/Group | Palbociclib With Aromatase Inhibitor
All-Cause Mortality (participants affected / at risk) | 62/242
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/47/NCT04394247/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/47/NCT04394247/SAP_001.pdf